CLINICAL TRIAL: NCT03174782
Title: Peripheral Nerve Blocks for Major Lower Extremity Amputations
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated due to not enough power and research staff assistance.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20107050
Record Dates: First submitted 2017-05-31; First posted 2017-06-05 (Actual); Results first posted 2023-05-31 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: To randomize patients, consent forms will be pre-labeled with a random subject identification number. This number will serve as the participants' study ID for all data collection in order to maintain privacy and confidentiality. Additionally, this number will be linked to a sealed envelope containing the random treatment group. The study coordinator will create the labels and assemble the envelopes to ensure all investigators remain blind to the treatment groups. This sealed envelope will be given to the anesthesia providers for the amputation. The anesthesia team will then administer the assigned treatment prior to induction of general anesthesia. Half of the patients will be randomized into the treatment group, and half of the patients will be randomized into the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment (Active Comparator): Patients randomized to the treatment group will receive regional nerve blocks (sciatic and femoral) with bupivacaine at the dose of 1 mg/kg.
  Interventions: Drug: Bupivacaine
- Control (Placebo Comparator): Patients randomized to the control group will receive two needle sticks (in the sciatic and femoral distributions) with normal saline to maintain the double-blinded investigation.
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Bupivacaine — Patients randomized to the treatment group will receive regional nerve blocks (sciatic and femoral) with bupivacaine at the dose of 1 mg/kg.
  Arms: Treatment
Drug: Saline Solution — Patients randomized to the control group will receive two needle sticks (in the sciatic and femoral distributions) with normal saline to maintain the double-blinded investigation.
  Arms: Control

SUMMARY:
This study will be a double-blinded randomized controlled trial analyzing all patients who will undergo major lower extremity amputations by the vascular surgery service at University of California, San Francisco (UCSF) Fresno between July 2017 and June 2018 to determine if regional nerve blocks (sciatic and femoral) have any effect on postoperative pain control, narcotic requirements, and length of stay compared with standard post-operative narcotic regimens.

DETAILED DESCRIPTION:
Major lower extremity amputations (above knee amputation or below knee amputation) are common procedures performed for patients with end stage ischemia, infection, and/or disfiguration. Patients undergoing major lower extremity amputations have significant morbidity and mortality. Up to 95% of amputees report chronic pain, and inadequate pre- and postoperative pain control may increase the risk of chronic amputation pain. Additionally, there is a growing epidemic of narcotic overdoses in the United States. From 2000 to 2014, the age-adjusted drug overdose death rate has more than doubled from 6.2 per 100,000 persons to 14.7 per 100,000. The main drugs associated with overdose deaths are prescription pain medications.

Regional nerve block is part of usual care and may serve as adjuncts for pain control after major lower extremity amputations. This pain control may be achieved by injecting bupivacaine into the sciatic and femoral nerves. Bupivacaine is an amide-type local anesthetic approved by the Food and Drug Administration (FDA) for local or regional anesthesia or analgesia for surgery. The dosage approved by the FDA for peripheral nerve blocks are 0.25% and 0.5%. The potential risks are central nervous system and cardiovascular system reactions. The central nervous system reactions are characterized by restlessness, anxiety, dizziness, or tremors. The cardiovascular system reactions are characterized by decreased cardiac output, heart block, hypotension, bradycardia, or arrhythmia. These risks are small and can be minimized further by slow administration and aspiration prior to administration to avoid intravascular injection. Other rare but potential risks of regional nerve block are nerve injury and hematoma formation.

Although bupivacaine is widely used for pain control, there are very few studies looking at regional nerve blocks as adjuncts for pain control after major lower extremity amputations. The number of randomized controlled trials is even fewer and none have been conducted in the United States. Baddoo looked at ten patients undergoing major lower extremity amputations (nine above knee amputations and one below knee amputation) with regional nerve blocks (a sciatic nerve block combined with either a 3-in-1 block or a psoas compartment lumbar plexus block). All ten patients were hemodynamically stable throughout surgery. Seven patients had good block, and three patients had fair block. Bech et al. presented a case report of four patients with severe cardiac insufficiency where they successfully utilized peripheral nerve blocks for trans-femoral amputation. The first patient was an 88-year-old man with American Society of Anesthesiologists (ASA) class 4. His echocardiogram showed an ejection fraction of 10%, mitral valve insufficiency and aortic valve sclerosis. The second patient was a 90-year-old woman with ASA class 4. Her echocardiogram showed an ejection fraction of 25% and severe mitral valve insufficiency. The third patient was a 64-year-old man with ASA class 4. His echocardiogram showed an ejection fraction of 25%, mitral valve insufficiency and tricuspid valve insufficiency. The fourth patient was a 74-year-old man with ASA class 4. His echocardiogram showed an ejection fraction of 15%, right-sided heart failure and both mitral and aortic valve insufficiency. All patients had successful outcomes in the postoperative course. Palkhiwala et al. looked at combined femoral and sciatic nerve blocks for lower limb procedures. With a randomized study involving 50 patients, they concluded that combined femoral and sciatic nerve blocks are effective for pain control with very low incidence of side effects. Forty-six out of fifty patients had complete block, and none of the patients had any cardiovascular or neurologic adverse events. Our study design is one of the first randomized controlled trials that looks at the effect of regional nerve blocks on postoperative pain and length of hospital stay.

This study will be a double-blinded randomized controlled trial analyzing patients undergoing major lower extremity amputation by the vascular surgery service at UCSF Fresno between July 2017 and June 2018 at Community Regional Medical Center, Clovis Community Medical Center, and Fresno Heart and Surgical Hospital. All patients who have been evaluated by the vascular surgery service and have had lower extremity amputation deemed necessary based on ischemic disease, infectious disease, and/or disfiguration will be included. Patients will be excluded if they are less than 18 years of age, pregnant, undergoing emergency amputations, staged amputations, or amputations by non-vascular surgeons, have known allergies to bupivacaine, are unable to communicate symptoms of pain, or refuse to participate in the study. Eligible patients may be identified by the vascular surgery service in their private office or following a consultation by the vascular surgery service in the hospital. Upon identification, eligible patients or their surrogate decision maker will be approached for consent by a member of the study team.

To randomize patients, consent forms will be pre-labeled with a random subject identification number. This number will serve as the participants' study identification (ID) for all data collection in order to maintain privacy and confidentiality. Additionally, this number will be linked to a sealed envelope containing the random treatment group. The study coordinator will create the labels and assemble the envelopes to ensure all investigators remain blind to the treatment groups. This sealed envelope will be given to the anesthesia providers for the amputation. The anesthesia team will then administer the assigned treatment prior to induction of general anesthesia. Half of the patients will be randomized into the treatment group, and half of the patients will be randomized into the control group.

Patients randomized to the treatment group will receive regional nerve blocks (sciatic and femoral) with bupivacaine at the dose of 1 mg/kg. The anesthesiologists are experts in pain management, and they are trained to perform regional nerve blocks. Femoral and sciatic nerve blocks are within their scope of practice, and they have been performing them quite frequently especially in orthopedic operations. Patients randomized to the control group will receive two needle sticks (in the sciatic and femoral distributions) with normal saline to maintain the double-blinded investigation. The anesthesiologists are not blinded in this study, and they will be able to provide the appropriate billing for the saline and the bupivacaine injections.

The remainder of the operation and post-operative course will proceed per the standard of care. Post-operative pain will be evaluated daily until discharge by the vascular surgery service using the McGill pain questionnaire. Additional data collected will include age, gender, race, BMI, ASA class, length of operation, hospital length of stay, oral and parenteral narcotic pain requirements. Any adverse events will immediately be reported to the Principal Investigator (PI) and the Institutional Review Board (IRB). A Medical Monitor with suitable expertise will be provided with all the study data on a monthly basis. The medical monitor will use that data especially the unforeseen adverse events and complications to ensure the study safety. The patients will be monitored and the data will be collected until six months after discharge.

ELIGIBILITY:
Inclusion Criteria:

* patients who require major lower extremity amputations

Exclusion Criteria:

* less than 18 years old, pregnant, emergency amputation, staged amputation, amputations performed by non-vascular surgeons, patients who are allergic to bupivacaine, patients who are unable to communicate symptoms of pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kamell Eckroth-Bernard, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Community Regional Medical Center, Fresno, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients included were evaluated by the vascular surgery service and had lower extremity amputation deemed necessary based on ischemic disease, infectious disease, and/or disfiguration. Patients were selected from 2018-2020 at the following sites; Community Regional Medical Center, Clovis Community Medical Center, and Fresno Heart and Surgical Hospital.
Period: Overall Study
Arm/Group | Treatment | Control
Started | 19 | 23
Completed | 18 | 22
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Unable to perform procedure by medical staff | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (14) | 58 (12) | 59 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 13 | 16 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 1 | 1 | 2
  Race: Hispanic | 7 | 13 | 20
  Race: White | 10 | 8 | 18
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28 (8) | 29 (6) | 29 (7)
Weight [Mean (Standard Deviation); unit: kg] | 80 (26) | 87 (20) | 84 (23)
Reason [Number; unit: participants]
  Ischemia | 10 | 7 | 15
  Infection | 2 | 5 | 7
  Wound | 2 | 5 | 7
  Osteomyelitis/ Charcot | 2 | 3 | 5
  Gangrene | 2 | 1 | 3
  Other | 1 | 2 | 3
Co-morbidities [Number; unit: participants]
  Hypertension (HTN) | 15 | 21 | 36
  Hyperlipidemia (HLD) | 6 | 14 | 20
  Diabetes Mellitus (DM) | 11 | 19 | 30
  Congestive Heart Failure (CHF) | 2 | 7 | 9
  End Stage Renal Disease (ESRD) | 5 | 3 | 8
  Peripheral Artery/Venous Disease | 4 | 10 | 14
  Coronary Artery Disease(CAD) | 3 | 6 | 9
  Smoker | 13 | 14 | 27
Laterality [Count of Participants; unit: Participants]
  Left | 9 | 10 | 19
  Right | 9 | 12 | 21

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain
Description: Postoperative pain will be assessed by McGill questionaire
Time Frame: 6 months
Population: No data were collected for this outcome measure since the study was terminated before collecting the outcome measure data.
Arm/Group | Treatment | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: No data were collected for All-Cause Mortality and Other (Not Including Serious) Adverse Events since the study was terminated before collecting this adverse event data.
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 6/18 | 3/22
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=18) | Control (N=22)
Complication (Injury, poisoning and procedural complications) | 6 | 3 — Postop complication include wound dehiscence and sternal wound infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT03174782/Prot_SAP_000.pdf